CLINICAL TRIAL: NCT05220891
Title: Comparison of Crystalloid and Colloid I.V Fluid Therapy in Prevention of Paracentesis Induced Circulatory Dysfunction (PICD) and Renal Dysfunction in Patients With Decompensated Liver Cirrhosis in Egypt: a Randomized Piolet Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shady Ashraf Kassem (Other)
Responsible Party: Sponsor-Investigator, Shady Ashraf Kassem, Resident, Assiut University
Organization: Assiut University (Other)
Other Study IDs: Ascitis control
Record Dates: First submitted 2022-01-15; First posted 2022-02-02 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Ascites
MeSH Terms: conditions — Ascites | interventions — Paracentesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Crystalloid group: Group( 1)Patients will be randomly assigned to be treated with crystalloid (n=30). They will receive an intravenous infusion of saline at a constant rate utilizing a pump infusion device (170 mL of 3.5% saline solution per liter of ascites removed at 999 mL/h). The amount of liquid infused and rate of infusion was selected based on previous studies (Sola-vera et al.,2003) Group (2)Patients will be randomly assigned to be treated with colloid (n=30). Albumin will be given at a dose of 8 g/L of ascitic fluid removed and will be infused immediately during the process of paracentesis.
  After paracentesis, diuretics and plasma expanders will be withheld until hospital discharge.
  Interventions: Other: Paracentesis
- Colloid group: Group (2)Patients will be randomly assigned to be treated with colloid (n=30). Albumin will be given at a dose of 8 g/L of ascitic fluid removed and will be infused immediately during the process of paracentesis.
  After paracentesis, diuretics and plasma expanders will be withheld until hospital discharge.
  Interventions: Other: Paracentesis

INTERVENTIONS:
Other: Paracentesis — Paracentesis from ascitic patient

SUMMARY:
2.2 Aim(s) of the Research (50 words max):

To Compare between crystalloid and colloid I.V fluid therapy in the prevention of paracentesis induced circulatory dysfunction (PICD) and renal dysfunction in patients with decompensated liver cirrhosis in Egypt.

To evaluate systemic vascular resistance in cirrhotic patients with tense ascites before and after therapeutic paracentesis.

DETAILED DESCRIPTION:
Background (Research Question, Available Data from the literature, Current strategy for dealing with the problem, Rationale of the research that paves the way to the aim(s) of the work). (200-250 words max.)

In the advanced stages of cirrhosis, there is pronounced arterial vasodilatation that further worsens by therapeutic paracentesis which plays a major role in causing circulatory dysfunction (El-Motey et al. 2013). Paracentesis-induced circulatory dysfunction (PICD) in cirrhotics with tense ascites develops in the majority of patients not receiving plasma volume expansion (Hamdy et al.,2014). Paracentesis induced circulatory dysfunction (PICD) will induce pronounced arterial vasodilatation in cirrhotic patients with tense ascites which can be prevented by the infusion of albumin, (Arora et al.,2020). albumin infusion is highly effective in preventing this disorder. However, albumin substitution is costly and holds the theoretical risk of infectious complications and allergic reactions (Arora et al.,2020). Various vasoconstrictors have also been used to prevent PICD such as terlipressin and noradrenaline. However, terlipressin is expensive and not available in some countries, and the use of noradrenaline requires intravenous (IV) infusion and intense monitoring (Singh et al .,2006), but there are few studies about the usage of crystalloids (Arora et al.,2020).

ELIGIBILITY:
Inclusion Criteria:

* Patients less than 70 years of age and more than 18 years, diagnosed as having liver cirrhosis with tense refractory ascites (> 5 liters). These diagnoses are determined by clinical, biochemical, morphological, and sonographic criteria.

Exclusion Criteria:

* Patients with blood pressure < 90/60 mmHg, and or HR > 110 b/m Patients with heart disease, pulmonary disease, alcohol consumption, pregnancy, hepatorenal syndrome Patients with hepatic encephalopathy, hepatorenal syndrome, or recent GIT haemorrage in last week Patients with spontaneous bacterial peritonitis or sepsis. Prothrombin time less than 30%, platelet count less than 30,000/mm3, serum creatinine level greater than 240 mmol/l Patients receiving any drugs that could interfere with cardiovascular, hepatic, or renal function, however, the use of diuretics and/or beta-blockers were permitted, but they were temporarily discontinued for 2 days before the investigations to eliminate the pharmacological influence on systemic vascular resistance work or volume status

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be randomly divided into two groups:
  Group( 1)Patients will be randomly assigned to be treated with crystalloid (n=30). They will receive an intravenous infusion of saline at a constant rate utilizing a pump infusion device (170 mL of 3.5% saline solution per liter of ascites removed at 999 mL/h). The amount of liquid infused and rate of infusion was selected based on previous studies (Sola-vera et al.,2003) Group (2)Patients will be randomly assigned to be treated with colloid (n=30). Albumin will be given at a dose of 8 g/L of ascitic fluid removed and will be infused immediately during the process of paracentesis.
  After paracentesis, diuretics and plasma expanders will be withheld until hospital discharge.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-01-11 (Estimated); Primary Completion 2024-01-11 (Estimated); Study Completion 2024-02-11 (Estimated)

PRIMARY OUTCOMES:
Paracentesis enduced circulatory dysfunction | Baseline
  The primary endpoint will be taken as the development of PICD. PICD will be defined as a significant drop in systemic vascular resistance before and after paracentesis using paired t-test with P-value < 0.05.

SECONDARY OUTCOMES:
Paracentesis induced renal impairment | Baseline
  Secondary (subsidiary):
  The secondary endpoint will be taken as the development of renal impairment or hyponatremia. Renal impairment will be defined as an increase in serum creatinine before and after paracentesis using paired t-test with P-value < 0.05. Hyponatremia is defined as a decrease in serum sodium >5mEq/L, to a level <130 mEq/L; in patients with a serum sodium concentration of <130 mEq/ L before treatment, hyponatremia will be defined as a decrease in serum sodium of >5mEq/L after paracentesi

REFERENCES:
- [Background] Arora V, Vijayaraghavan R, Maiwall R, Sahney A, Thomas SS, Ali R, Jain P, Kumar G, Sarin SK. Paracentesis-Induced Circulatory Dysfunction With Modest-Volume Paracentesis Is Partly Ameliorated by Albumin Infusion in Acute-on-Chronic Liver Failure. Hepatology. 2020 Sep;72(3):1043-1055. doi: 10.1002/hep.31071. Epub 2020 Jul 9. PMID 31849085
- [Background] Darnis E, Boysen S, Merveille AC, Desquilbet L, Chalhoub S, Gommeren K. Establishment of reference values of the caudal vena cava by fast-ultrasonography through different views in healthy dogs. J Vet Intern Med. 2018 Jul;32(4):1308-1318. doi: 10.1111/jvim.15136. Epub 2018 May 10. PMID 29749656
- [Background] Richert A, Raines D, Lopez FA. New onset ascites secondary to cirrhosis. J La State Med Soc. 2009 Jan-Feb;161(1):9-13; quiz 13, 54. No abstract available. PMID 19278163
- [Background] Moller S, Henriksen JH, Bendtsen F. Ascites: pathogenesis and therapeutic principles. Scand J Gastroenterol. 2009;44(8):902-11. doi: 10.1080/00365520902912555. PMID 19479632
- [Background] Novo Matos J, Pereira N, Glaus T, Wilkie L, Borgeat K, Loureiro J, Silva J, Law V, Kranjc A, Connolly DJ, Luis Fuentes V. Transient Myocardial Thickening in Cats Associated with Heart Failure. J Vet Intern Med. 2018 Jan;32(1):48-56. doi: 10.1111/jvim.14897. Epub 2017 Dec 15. PMID 29243322
- [Background] Marwick TH, Gillebert TC, Aurigemma G, Chirinos J, Derumeaux G, Galderisi M, Gottdiener J, Haluska B, Ofili E, Segers P, Senior R, Tapp RJ, Zamorano JL. Recommendations on the use of echocardiography in adult hypertension: a report from the European Association of Cardiovascular Imaging (EACVI) and the American Society of Echocardiography (ASE)dagger. Eur Heart J Cardiovasc Imaging. 2015 Jun;16(6):577-605. doi: 10.1093/ehjci/jev076. PMID 25995329
- [Background] Singh V, Kumar R, Nain CK, Singh B, Sharma AK. Terlipressin versus albumin in paracentesis-induced circulatory dysfunction in cirrhosis: a randomized study. J Gastroenterol Hepatol. 2006 Jan;21(1 Pt 2):303-7. doi: 10.1111/j.1440-1746.2006.04182.x. PMID 16460491
- [Background] Shah AM, Cikes M, Prasad N, Li G, Getchevski S, Claggett B, Rizkala A, Lukashevich I, O'Meara E, Ryan JJ, Shah SJ, Mullens W, Zile MR, Lam CSP, McMurray JJV, Solomon SD; PARAGON-HF Investigators. Echocardiographic Features of Patients With Heart Failure and Preserved Left Ventricular Ejection Fraction. J Am Coll Cardiol. 2019 Dec 10;74(23):2858-2873. doi: 10.1016/j.jacc.2019.09.063. PMID 31806129
- [Background] Runyon BA; AASLD Practice Guidelines Committee. Management of adult patients with ascites due to cirrhosis: an update. Hepatology. 2009 Jun;49(6):2087-107. doi: 10.1002/hep.22853. No abstract available. PMID 19475696
- [Background] Sola-Vera J, Minana J, Ricart E, Planella M, Gonzalez B, Torras X, Rodriguez J, Such J, Pascual S, Soriano G, Perez-Mateo M, Guarner C. Randomized trial comparing albumin and saline in the prevention of paracentesis-induced circulatory dysfunction in cirrhotic patients with ascites. Hepatology. 2003 May;37(5):1147-53. doi: 10.1053/jhep.2003.50169. PMID 12717396